CLINICAL TRIAL: NCT04159012
Title: NESBID: Neuro-Stimulation of the Brain in Depression. A Randomized, Controlled Clinical Trial of Transcranial Direct Current Stimulation Augmentation, as Compared to Sham Therapy, in the Treatment of Ultra-resistant Major Depressive Disorder
Brief Title: NESBID: Neuro-Stimulation of the Brain in Depression
Acronym: NESBID
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Logistical reasons
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TDCS2019
Record Dates: First submitted 2019-07-08; First posted 2019-11-12 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Transcranial Direct Current Stimulation; Electric Stimulation Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active transcranial direct current stimulation (Experimental): Active transcranial direct current stimulation (tDCS), delivered at 2 mA and for 30 minutes, on sequential weekdays, for a total of 30 sessions. Participants will continue to receive their usual pharmacotherapy and psychotherapy.
  Interventions: Device: Transcranial direct current stimulation
- Sham transcranial direct current stimulation (Sham Comparator): Sham transcranial direct current stimulation (tDCS), which will ramp up to 2 mA over 17 s, and then ramp down to and remain at 0.3 mA for the remainder of the 30 minute session. The short period of active stimulation is included to stimulate the somatic sensations of active therapy. The trickle current at 0.3 mA is necessary to measure electrode contact and prevent investigators from deducing that the device is no longer active. Participants will receive the sham therapy on sequential weekdays for a total of 30 sessions. Participants will continue to receive their usual pharmacotherapy and psychotherapy.
  Interventions: Device: Transcranial direct current stimulation

INTERVENTIONS:
Device: Transcranial direct current stimulation — A Sooma transcranial direct current stimulator, using carbon electrodes, a reusable cap (to promote reproducible electrode placement), and disposable sponges that will be soaked in normal saline.
  The anode will be positioned over the left dorsolateral prefrontal cortex (position F3 on the 10-20 the International EEG system), and the cathode will be positioned over the right dorsolateral prefrontal cortex (position F4).
  Other Names: Sooma tDCS

SUMMARY:
In Canada, approximately 20% of patients with Major Depressive Disorder (MDD) have treatment-resistance and fail to respond to trials of pharmacotherapy or psychotherapy. Although the treatment of choice has historically consisted of electroconvulsive therapy (ECT), this is not always feasible or practical, and carries a risk of side-effects that may be unacceptable to certain patients.

In this pragmatic, multi-site, placebo-controlled and double-blinded clinical trial, participants with ultra treatment-resistant MDD will be randomized to receive either active or sham transcranial direct current stimulation in addition to their usual treatment. Ultra treatment-resistant depression will be operationally defined as MDD that has failed to respond to at least five previous trials of antidepressants at sufficient doses, or ECT, or ketamine. Patients will receive a total of 30 active or sham treatment sessions (5 per week), for 30 minutes per session. In both groups, the anode will be placed over the left dorsolateral prefrontal cortex (position F3), and the cathode over the right dorsolateral prefrontal cortex (position F4). Patients in the sham group will receive electrical stimulation at 2 mA for less than 30 seconds, whereas patients in the active group will receive that level of stimulation for the entire duration of treatment.

The study's primary outcome is the change in score on a clinician-graded depression inventory (the Montgomery-Asberg Depression Rating Scales). Secondary outcomes include change in scores on a self-administered depression rating scale and measurement of function scale. Information on language ability will also be collected, as will data on side-effects of treatment. Scores will be collected before the trial start, after every 10 sessions, and one month after trial completion.

ELIGIBILITY:
Inclusion Criteria:

* Currently suffering from an MDE with a score on the Montgomery-Åsberg Depression Rating Scale (MADRS) greater than 34 (signifying severe depression)
* Have ultra treatment resistant MDD (defined as failure to remit despite adequate trials with five antidepressants, or failure to remit with ECT, or failure to remit with ketamine)

Exclusion Criteria:

* Have been diagnosed with psychosis, an addiction disorder (other than nicotine), borderline personality disorder, or antisocial personality disorder, as these conditions could interfere with adherence to the study protocol
* Are currently using a herbal compound or known NMDA-modulating agent, as these substances could interfere with the induction of LTP and thereby limit the effectiveness of tDCS
* Are pregnant, as tDCS has not been adequately studied in this population
* Have an electronic implant, cardiac dysrhythmia, seizure disorder, neurological disorder, or neurosurgical history, as the safety of electrical stimulation with tDCS cannot be assured given these comorbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Baseline, after 2 weeks, after 4 weeks, after 6 weeks/trial completion, and 1 month after trial completion
  An observer-assessed score of depression severity. The total is scored from 0 to 60, with higher scores representing greater depression severity

SECONDARY OUTCOMES:
Quick Inventory of Depressive Symptomatology - Self Report (QIDS-SR16) | Baseline, after 2 weeks, after 4 weeks, after 6 weeks/trial completion, and 1 month after trial completion
  A participant-assessed measurement of depression severity. The total is scored from 0 to 27, with higher scores indicating greater depression severity.
World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0) | Baseline, after 2 weeks, after 4 weeks, after 6 weeks/trial completion, and 1 month after trial completion
  Change in the World Health Organization Disability Assessment Schedule score
Exploratory language analysis | Baseline and after 6 weeks/trial completion
  Change in language characteristics, based on recorded interviews
Lexical decision making task | Baseline and after 6 weeks/trial completion
  Performance on a task in which patients much distinguish real from fictitious words as quickly as possible
tDCS adverse events scale | Baseline, after 2 weeks, after 4 weeks, after 6 weeks/trial completion, and 1 month after trial completion
  Adverse events as assessed on a scale derived from a systematic review on side effects that may be associated with tDCS
FIBSER | Baseline, after 2 weeks, after 4 weeks, after 6 weeks/trial completion, and 1 month after trial completion
  Frequency, Intensity, and Burden of Side-Effects Rating Scale
PRISE | Baseline, after 2 weeks, after 4 weeks, after 6 weeks/trial completion, and 1 month after trial completion
  Patient-Rated Inventory of Side-Effects Scale
YMRS | Baseline, after 2 weeks, after 4 weeks, after 6 weeks/trial completion, and 1 month after trial completion
  Young Mania Rating Scale, included to capture treatment-related manic or hypomanic switches

CONTACTS AND LOCATIONS:
Overall Officials: Serdar M Dursun, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- Grey Nuns Community Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.

REFERENCES:
- [Derived] Suleman R, Tucker BV, Dursun SM, Demas ML. The Neurostimulation of the Brain in Depression Trial: Protocol for a Randomized Controlled Trial of Transcranial Direct Current Stimulation in Treatment-Resistant Depression. JMIR Res Protoc. 2021 Mar 17;10(3):e22805. doi: 10.2196/22805. PMID 33729165